CLINICAL TRIAL: NCT04736719
Title: Replication of the AMPLIFY Anticoagulant Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-AMPLIFY
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Warfarin: Reference group
  Interventions: Drug: Warfarin
- Apixaban: Exposure group
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Apixaban dispensing claim is used as the exposure group
  Groups: Apixaban
Drug: Warfarin — Warfarin dispensing claim is used as the reference group
  Groups: Warfarin

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates through standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates:

Market availability of apixaban in the U.S. for treatment of deep vein thrombosis and pulmonary embolism started on August 21, 2014.

* For Medicare: August 21, 2014 - December 31, 2017 (end of available data)
* For Marketscan: August 21, 2014 - December 31, 2018 (end of available data)
* For Optum: August 21, 2014 - March 31, 2020 (end of available data)

Inclusion Criteria:

* Either:

  * Acute symptomatic proximal deep vein thrombosis (DVT) with evidence of proximal thrombosis that involves at least the popliteal vein or a more proximal vein, demonstrated by imaging with: compression ultrasound (CUS), including grey-scale or color-coded Doppler, OR - ascending contrast venography
  * Acute symptomatic PE with evidence of thrombosis demonstrated by imaging as follows:

    1. an intraluminal filling defect in segmental or more proximal branches on spiral computed tomography (CT) scan
    2. an intraluminal filling defect or a sudden cutoff of vessels more than 2.5 mm in diameter on the pulmonary angiogram
    3. a perfusion defect of at least 75% of a segment with a local normal ventilation result (high probability) on ventilation/perfusion lung scan (VPLS)
* Men and women ages 18 years or greater

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method of birth control (such as oral contraceptives, other hormonal contraceptives [vaginal products, skin patches, or implanted or injectable products], or mechanical products such as an intrauterine device or barrier methods [diaphragm, condoms, spermicides]) to avoid pregnancy for the entire study
* Women who are pregnant or breast feeding
* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of venous thromboembolism (VTE)
* Active bleeding or high risk for bleeding contraindicating treatment with low-molecular weight heparin (LMWH) and a vitamin K antagonist (VKA)
* Presence of a mechanical valve
* Intracranial bleeding, intraocular bleeding, gastrointestinal bleeding 6 months prior to enrollment date
* Head trauma or other major trauma 2 months prior to enrollment date
* Ischemic stroke or neurosurgery 1 week prior to enrollment date
* Any of the following one day prior to and including date of enrollment:

  * Gross hematuria
  * Evidence of poor healing of a major wound
  * Intracranial neoplasm, arteriovenous malformation or aneurysm
  * Overt major bleeding
  * Documented hemorrhagic tendencies or blood dyscrasias
* Any of the following 6 months prior to or on the day of enrollment:

  * Active and clinically significant liver disease
  * Life expectancy < 6 months
  * Bacterial endocarditis
  * Uncontrolled hypertension: systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg; (subjects who have a transient, higher blood pressure elevation associated with acute PE [upper limit: systolic blood pressure 200 mm Hg or diastolic blood pressure 100 mm Hg] may enter the study;) elevated blood pressure that is persistent 1-2 days after the index DVT or PE should be treated according to local guidelines
  * Platelet count <100,000/mm3
  * Hemoglobin <9 g/dL
  * Serum creatinine >2.5 mg/dL (221 umol/L)
  * Calculated creatinine clearance <25 ml/min
  * ALT or AST >2 times upper limit of normal
  * Total bilirubin >1.5 times upper limit of normal (unless an alternative causative factor is identified [eg, Gilbert's syndrome])
  * Heparin-induced thrombocytopenia
* Subjects requiring aspirin (ASA) >165 mg/day on day prior to or on day of enrollment
* Subjects requiring dual antiplatelet therapy (ASA plus clopidogrel or ASA plus ticlopidine) one day prior to or on enrollment. Subjects who transition from dual antiplatelet therapy to monotherapy prior to randomization will be eligible for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing apixaban to warfarin users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of apixaban or warfarin (index date). We will restrict the analyses to patients with a diagnosis of proximal DVT, PE, or both.
Sampling Method: Non-Probability Sample
Enrollment: 19002 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with composite of VTE and VTE-related mortality | Through study completion (a median of 74 - 96 days)

SECONDARY OUTCOMES:
Number of patients with hospital admission for VTE | Through study completion (a median of 74 - 96 days)
Number of patients with VTE-related mortality | Through study completion ( a median of 74-96 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT04736719/Prot_SAP_001.pdf